CLINICAL TRIAL: NCT06345508
Title: Quantitative Ultrasound to Improve Detection and Diagnosis of Liver Cancer
Brief Title: Early Detection of Liver Cancer by QUS
Acronym: QUS in HCC
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-12161
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Ultrasound; Quantitative ultrasound (QUS); Liver cancer; Hepatocellular carcinoma; Elastography; Viscoelastography; Screening; Surveillance; Diagnosis; Diagnostic performance
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantitative Ultrasound — Research quantitative ultrasound
  Other Names: QUS
Diagnostic Test: B-mode Ultrasound — B-mode US performed according to the clinical standard of care.
  Other Names: B-mode US
Diagnostic Test: Magnetic Resonance Imaging — The composite reference standard includes MRI performed according to the clinical standard of care or histopathology when available.
  Other Names: MRI
Diagnostic Test: Liver Biopsy — The composite reference standard includes MRI performed according to the clinical standard of care or histopathology when available.

SUMMARY:
Worldwide, liver cancers are the third most common cause of cancer mortality. Even when liver cancer is suspected by blood tests, imaging is required to determine the location, size, and extent of disease. Medical societies therefore recommend surveillance with ultrasound every 6 months in at-risk patients. However, a key challenge to improving the survival is that ultrasound may miss half of early-stage liver cancers, thus diagnosis must rely on additional tests such as computed tomography (CT), magnetic resonance imaging (MRI), or biopsy. Hence, there is a clear need to improve the ability to detect liver cancers, especially with ultrasound. The investigator's team proposes novel ultrasound approaches to detect cancer nodules invisible on conventional ultrasound based on differences in mechanical and structural properties between liver and tumor. Improving detection is critical because liver cancer can be cured only if detected at an early stage, as shown by improvements in survival rates in patients enrolled in surveillance programs. The investigator's multi-disciplinary, national, and international team includes experts in clinical fields (hepatology, oncology, radiology, pathology), basic sciences (engineering, medical physics, machine learning, biostatistics), and patient partnership. The investirgator will apply the methodology of patient partner recruitment and collaborate with the Centre of Excellence on Partnership with Patients and the Public to select potential new collaborators. This will permit this project to be informed at every stage by patient and family perspectives, ensuring that the results of this project will be more robust, impactful, and aligned with the priorities, needs and experiences of those who live with liver cancer. The investigator submits a research proposal focused on advanced imaging techniques because imaging constitutes a foundation for surveillance, diagnosis, staging, treatment selection and assessment of treatment response in patients with liver cancer.

DETAILED DESCRIPTION:
BACKGROUND Worldwide, liver cancers are the third most common cause of cancer mortality. In Canada, hepatocellular carcinoma (HCC) is one of the few cancers for which mortality is increasing. Early detection of HCC improves the likelihood of curative treatment and survival. Systematic HCC surveillance with ultrasound (US) is recommended by practice guidelines. However, conventional (B-mode) US suffers from low sensitivity (47%) for detecting early-stage HCC due to fatty liver, obesity, and cirrhosis. Once a suspicious nodule is detected by US, guidelines recommend contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) to confirm cancer. Hence, there is an urgent need to improve the ability to detect and diagnose HCC early. Members of the investigator's team have developed innovative quantitative ultrasound (QUS) techniques (including shear wave viscoelastography [SWV] and sub-resolution cellular imaging) that have a high diagnostic potential. The investirgator hypothesizes that a combination of QUS techniques offering complementary assessment of tissue characteristics will improve our ability to detect liver nodules and diagnose HCC.

METHODOLOGY Design: Prospective, cross-sectional imaging trial comparing head-to-head B-mode US and research QUS acquired within one month to the composite reference standard. Reference standard: MRI will be used as the non-invasive ground truth for liver nodules detection and classification except when biopsy is available. Data analysis: Lesion detectability will be measured by contrast-to-noise ratio on US and QUS maps for different size thresholds (<10 mm, 10-20 mm, >20 mm) used in diagnostic algorithms. Diagnostic performance will be measured by receiver operating characteristic curve analysis on the training and test sets for different size thresholds. The diagnostic accuracy of US and QUS + B-mode US will be compared by using the DeLong method.

RATIONALE AND IMPACT Early detection through systematic US surveillance translates into curative therapy in a higher proportion of patients and into improvements in survival rates. This imaging trial will provide a low-cost imaging technique to identify liver cancers earlier and from a single exam. Unlike some other imaging techniques, US is widely available throughout Canada. A major impact of this work, for patients and medical institutions, will be to lower the need for liver biopsy, the risk of complications and the cost for HCC diagnosis. This trial will position Canada as a leader in HCC diagnosis as new QUS and SWV biomarkers will be tested.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients scheduled for US- or MRI-based surveillance of HCC or undergoing MRI-based imaging for characterization of liver nodules as part of their clinical standard of care.

Exclusion Criteria:

- Patients with prior locoregional or systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for US- or MRI-based surveillance of HCC or undergoing MRI-based imaging for characterization of liver nodules as part of their clinical standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 328 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Compare the sensitivity of QUS + B-mode US vs B-mode US alone for lesion detection, using MRI as the reference standard for detection | Within one month of the composite reference test (conventional MRI or pathology).
  Lesion detectability will be measured by contrast-to-noise ratio on US and QUS maps for different size thresholds (<10 mm, 10-20 mm, >20 mm) used in diagnostic algorithms

SECONDARY OUTCOMES:
Compare the specificity of QUS + B-mode US vs B-mode US alone for diagnosis of HCC, using MRI or biopsy as the composite reference standard for classification | Within one month of the composite reference test (conventional MRI or pathology).
  Diagnostic performance will be measured by receiver operating characteristic curve analysis on the training and test sets for different size thresholds
Determine the lesion-to-liver contrast of investigational QUS techniques for detection of HCC | Within one month of the composite reference test (conventional MRI or pathology).
  The diagnostic accuracy of US and QUS + B-mode US will be compared by using the DeLong method

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada